CLINICAL TRIAL: NCT03005054
Title: Open-label, Controlled, Randomized, Multicenter, Dose Escalation Study Evaluating the Safety, Tolerability, and Efficacy of Single or Multiple Applications of StrataGraft® Skin Tissue as an Alternative to Autografting Full-thickness Complex Skin Defects
Brief Title: StrataGraft® Skin Tissue as an Alternative to Autografting Full-thickness Complex Skin Defects
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Protracted enrollment and limited wound closure in the first three subjects
Sponsor: Stratatech, a Mallinckrodt Company (Industry)
Responsible Party: Sponsor
Organization: Mallinckrodt (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STRATA2014; W81XWH-16-C-0202 (Other Grant/Funding Number: DoD)
Record Dates: First submitted 2016-12-21; First posted 2016-12-29 (Estimated); Results first posted 2021-08-03 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Trauma-related Wound; Burns; Skin Wound
Keywords: Full-thickness; Acute trauma
MeSH Terms: conditions — Burns | interventions — Transplantation, Autologous

STUDY DESIGN:
Intervention Model Description: See detailed description
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- StrataGraft skin tissue (Experimental)
  Interventions: Biological: StrataGraft Skin Tissue; Procedure: Autograft

INTERVENTIONS:
Biological: StrataGraft Skin Tissue — StrataGraft® skin tissue is provided as a suturable rectangular piece of stratified epithelial tissue composed of a living dermal matrix containing dermal fibroblasts overlaid with human epidermal keratinocytes (NIKS®).
Procedure: Autograft — The current standard of care procedure for the treatment of severe complex skin defects. The procedure involves the removal of a sheet of healthy skin from an uninjured site on the patient and using it to cover the original wound.

SUMMARY:
About 20 participants will be enrolled in this trial if they have had an accident that damages both the dermal (outside) and epidermal (inside) layers of skin on up to 49% of their body.

This condition is called full-thickness complex skin defects resulting from acute traumatic skin loss.

Participants will be treated with StrataGraft skin tissue to evaluate it's safety and effectiveness for use in treating full-thickness complex skin defects.

DETAILED DESCRIPTION:
The objective of this range-finding study was to assess the safety, tolerability, and efficacy of single or repeated application of StrataGraft skin tissue in full-thickness complex skin defects resulting from acute traumatic skin loss (eg, thermal burns or degloving injuries) requiring surgical excision and autografting.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18-65 years, inclusive
2. Written informed consent
3. Sufficient healthy skin identified and reserved as a donor site in the event that the StrataGraft treatment site requires autografting
4. Complex skin defects of up to 49% Total Body Surface Area (TBSA) requiring excision and autografting

   * Total skin defect may consist of more than one wound area
5. Full-thickness complex skin defects requiring excision and autografting
6. Study treatment sites on the torso and limbs may be up to 200 cm2 in cohort 1 and 400 cm2 in cohort 2
7. For thermal burns only, first excision and grafting of treatment sites

Exclusion Criteria:

1. Pregnant women and prisoners
2. Subjects receiving systemic immunosuppressive therapy
3. Subjects with a known history of malignancy
4. Preadmission insulin-dependent diabetic subjects
5. Subjects with concurrent conditions that in the opinion of the investigator may compromise subject safety or study objectives
6. Expected survival of less than three months
7. Participation in the treatment group of an interventional study within the 90 days prior to enrollment
8. Chronic wounds
9. The face, head, neck, hands, feet, buttocks, perineum, and area over joints
10. Treatment sites with exposed tendon or bony prominences
11. Chemical and electrical burns
12. Treatment sites adjacent to unexcised eschar
13. Clinical suspicion of infection at the anticipated treatment sites

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2019-03-26 (Actual); Study Completion 2019-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Mallinckrodt
Locations (4):
- United States (4):
  - Arizona Burn Center, Phoenix, Arizona
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - U.S. Army Institute of Surgical Research Adult Burn Center, Fort Sam Houston, Texas
  - University of Wisconsin Hospital, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No
Discussion of statistical endpoints and analysis are included in manuscripts. Summary aggregate (basic) results (including adverse events information) and the study protocol are made available on clinicaltrials.gov (NCT03005054) when required by regulation. Individual de-identified patient data will not be disclosed. Requests for additional information should be directed to the company at medinfo@mnk.com.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | StrataGraft Skin Tissue
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants
Arm/Group | StrataGraft Skin Tissue
Number analyzed (Participants) | 3
Age, Continuous [Median (Full Range); unit: years] | 53 [21 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White: Not Hispanic or Latino | 3
  White: Hispanic or Latino | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Percent Area of the StrataGraft Treatment Site Requiring Autografting by Three Months
Description: The percentage of the treatment site area initially covered with StrataGraft tissue that requires autograft by three months will be determined.
Time Frame: 3 months
Population: All participants
Measure: Number; unit: percentage of treatment site
Arm/Group | StrataGraft Skin Tissue
Number analyzed (Participants) | 3
percentage of treatment site
  Participant 1 | 100
  Participant 2 | 25
  Participant 3 | 125

2. Primary Outcome: Percentage of Participants With Complete Wound Closure of the Treatment Sites at Three Months
Description: Complete wound closure is defined as ≥95% re-epithelialization of all treatment sites with the absence of drainage
Time Frame: 3 months
Population: All participants
Measure: Number; unit: percentage of participants
Arm/Group | StrataGraft Skin Tissue
Number analyzed (Participants) | 3
percentage of participants | 100

3. Secondary Outcome: Percent of Subjects Requiring Autografting of the StrataGraft Treatment Site by 3 Months
Time Frame: within 3 months
Population: Data were not collected
Arm/Group | StrataGraft Skin Tissue
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Participants With Complete Wound Closure of the Treatment Sites at 3, 6, and 12 Months
Time Frame: within 3, 6 and 12 months
Population: Data were not collected
Arm/Group | StrataGraft Skin Tissue
Number analyzed (Participants) | 0

5. Secondary Outcome: Percent Wound Closure at 3, 6, and 12 Months
Time Frame: within 3, 6, and 12 Months
Population: Data were not collected
Arm/Group | StrataGraft Skin Tissue
Number analyzed (Participants) | 0

6. Secondary Outcome: Cosmesis of Treatment Sites at 3, 6, and 12 Months
Description: Cosmesis is defined as the preservation, restoration, or enhancement of physical appearance
Time Frame: within 3, 6, and 12 Months
Population: Data were not collected
Arm/Group | StrataGraft Skin Tissue
Number analyzed (Participants) | 0

7. Secondary Outcome: Cosmesis of Donor Sites at 3, 6, and 12 Months
Description: Cosmesis is defined as the preservation, restoration, or enhancement of physical appearance
Time Frame: within 3, 6, and 12 Months
Population: Data were not collected
Arm/Group | StrataGraft Skin Tissue
Number analyzed (Participants) | 0

8. Secondary Outcome: Pain of Donor Sites Measured at Days 3, 7, 14, 21, and 28
Time Frame: at days 3, 7, 14, 21, and 28
Population: Data were not collected
Arm/Group | StrataGraft Skin Tissue
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 3 months
Description: Tables reflect treatment-emergent adverse events (TEAEs). If a subject has more than one incidence of a preferred term, the subject is counted only once for that preferred term.
Arm/Group | StrataGraft Skin Tissue
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | StrataGraft Skin Tissue (N=3)
Graft complication (Injury, poisoning and procedural complications) | 1 — Unrelated to treatment
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | StrataGraft Skin Tissue (N=3)
Graft complication (Injury, poisoning and procedural complications) | 2
Fungal skin infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Hyperglycaemia (Endocrine disorders) | 1
Cataract (Eye disorders) | 1
Pain (General disorders) | 1
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Blister (Skin and subcutaneous tissue disorders) | 1
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
Due to protracted enrollment and limited wound closure in the first three subjects, the Sponsor decided to end further enrollment and the study was terminated with only 3 subjects enrolled into Cohort 1. No participants were enrolled into Cohort 2. Therefore, posted results include primary outcome measures for the 3 subjects enrolled, but no data for the secondary outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-23): https://cdn.clinicaltrials.gov/large-docs/54/NCT03005054/Prot_SAP_000.pdf